CLINICAL TRIAL: NCT02529033
Title: Comparative Hemodynamic Assessment Between Lidco Rapid and Pulmonary Artery Thermodilution
Brief Title: Hemodynamic Survey Cardiac Surgical Scenarios
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: 201504777
Record Dates: First submitted 2015-08-03; First posted 2015-08-19 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Low Cardiac Output
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: LIDCO Rapid, Pulmonary artery catheter — Hemodynamic monitoring systems

SUMMARY:
The purpose of this study is to find out the Lidco Rapid ( monitoring tool gives cardiac output) is as equivalent in determining the hemodynamic assessment in cardiac surgical scenarios as the most often used pulmonary artery catheter, which is much more invasive than the Lidco Rapid. This will be accomplished through online surveys which have different cardiac surgery scenarios and will be distributed to cardiac fellowship trained anesthesiologists. The online based survey will include a specific scenario and details on the scenario represented in image format and a brief description of the patient to aid with their analysis of the situation.

DETAILED DESCRIPTION:
Data from PA catheter such as PA pressure, pulmonary wedge pressure and cardiac output has been widely used in the various clinical situations warranting advance hemodynamic monitoring. It is considered as gold standard but unfortunately there is always risk associated with PA catheter and time lag between the clinical events and interpretation. Lidco Rapid is one of the non-invasive hemodynamic tools to measure various parameters. It is widely used in the intensive care set up for goal directed therapy but unfortunately there is not enough data to show whether it is useful in various peri-operative clinical conditions. In the online based survey, responses from the participants are recorded in the nominal scale ( 1 to 5 where 3 represents near normal). This survey will help to determine whether Investigators can replace the Lidco in any clinical situation warranting advance hemodynamic monitoring.

No previous study was done to specifically find out the hemodynamic component that differs between these tools intraoperatively in varying hemodynamic conditions during cardiac surgery although there were few studies compared the trend in the cardiac output with difference in opinion on their accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Must be a certified Anesthesiologist with cardiac fellowship training

Exclusion Criteria:

* none

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac Fellowship trained Anesthesiologists
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To expect difference is within 1 unit ( scale of 1 to 5) in the hemodynamic assessment preferably preload , afterload and contractility between Lidco and data from PA catheter in different cardiac surgical patient scenarios. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Subramani, M.D., Principal Investigator — University of Iowa

REFERENCES:
- [Background] Hadian M, Kim HK, Severyn DA, Pinsky MR. Cross-comparison of cardiac output trending accuracy of LiDCO, PiCCO, FloTrac and pulmonary artery catheters. Crit Care. 2010;14(6):R212. doi: 10.1186/cc9335. Epub 2010 Nov 23. PMID 21092290
- [Background] Broch O, Renner J, Hocker J, Gruenewald M, Meybohm P, Schottler J, Steinfath M, Bein B. Uncalibrated pulse power analysis fails to reliably measure cardiac output in patients undergoing coronary artery bypass surgery. Crit Care. 2011;15(1):R76. doi: 10.1186/cc10065. Epub 2011 Feb 28. PMID 21356060